CLINICAL TRIAL: NCT06342869
Title: Comparison of the Effects of Lidocaine and Articaine Used for Buccal Infiltration and Supplemental Palatinal Infiltration Anesthesia in Teeth With Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Damla Kırıcı, associate professor, Akdeniz University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 690
Record Dates: First submitted 2024-02-28; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Fist and Second Molars With ırreversible Pulpitis
Keywords: articaine, lidocaine, irreversible pulpitis, infiltration anesthesia
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- buccal infiltration with 4% articaine containing 1:100,000 epinephrine (Experimental)
  Interventions: Procedure: Anesthesia
- buccal infiltration with 2% lidocaine containing 80,000 epinephrine (Experimental)
  Interventions: Procedure: Anesthesia
- buccal and palatinal infiltration with 4% articaine containing 1:100,000 epinephrine (Experimental)
  Interventions: Procedure: Anesthesia
- buccal and palatinal infiltration with 2% lidocaine containing 80.000 epinephrine (Experimental)
  Interventions: Procedure: Anesthesia

INTERVENTIONS:
Procedure: Anesthesia — application of different anesthesia techniques

SUMMARY:
Objective: The aim of this study was to compare the effects of articaine or lidocaine in buccal infiltration or palatal infiltration in addition to buccal infiltration in maxillary first or second molars with irreversible pulpitis.

Method: Among the patients who applied to Akdeniz University Faculty of Dentistry Endodontic Clinic for the treatment of maxillary molars with irreversible pulpitis, 80 volunteers who met the criteria were included in the study. Eighty patients were divided into 4 groups (n = 20). 1. group buccal infiltration with 4% articaine containing 1:100,000 epinephrine, 2. group buccal infiltration with 2% lidocaine containing 80,000 epinephrine, 3. group buccal and palatinal infiltration with 4% articaine containing 1:100,000 epinephrine, 4.group buccal and palatinal infiltration with 2% lidocaine containing 80.000 epinephrine. Pain during the endodontic procedure was determined and recorded according to the Heft Parker visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be a healthy individual between the ages of 18 and 65 who is classified as ASA I and II.
2. No allergy to local anesthetic substances to be used in the study
3. Upper maxillary molars with irreversible pulpitis whose vitality has been proven by pulp tests, with no radiolucency at the root tip
4. Not having used any painkillers, antibiotics, antidepressants and sedative drugs in the last 12 hours
5. Being capable of understanding the Pain scale

Exclusion Criteria:

1. Allergy to local anesthetics
2. Failure to respond to the cold test and electric pulp test performed on the relevant tooth
3. Radiolucent lesion in the apical part of the relevant tooth on periapical radiography
4. No vital tissue is encountered when the pulp chamber is opened

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of complementary palatinal anesthesia with VAS | 10 minutes after anesthesia is performed

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kanaa MD, Whitworth JM, Meechan JG. A comparison of the efficacy of 4% articaine with 1:100,000 epinephrine and 2% lidocaine with 1:80,000 epinephrine in achieving pulpal anesthesia in maxillary teeth with irreversible pulpitis. J Endod. 2012 Mar;38(3):279-82. doi: 10.1016/j.joen.2011.11.010. Epub 2011 Dec 22. PMID 22341059
- [Derived] Kolay D, Kirici D. Comparison of the effects of lidocaine and articaine used for buccal infiltration and supplemental palatinal infiltration anesthesia in maxillary molars with irreversible pulpitis: a prospective randomized study. BMC Oral Health. 2025 Feb 8;25(1):207. doi: 10.1186/s12903-025-05552-y. PMID 39923048